CLINICAL TRIAL: NCT01970761
Title: Alleviation of Neuropathic Scar Pain With Autologous Fat Graft
Brief Title: Autologous Fat Graft Alleviate Scar Pain
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUH-IRB-20120246
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2012-12

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- scar, Fat Graft, Visual Analogue Scale: patients received autologous fat grafting in scar areas

SUMMARY:
Traumatic wounds inflict small- and large-fiber sensory nerve damage, causing neuropathic pain in scar tissue. Autologous fat grafting has been clinically shown to improve scar quality, but scantly study has explored its effects on pain. The aim of the study was to survey its effect on pain.

DETAILED DESCRIPTION:
Methods: From February 2008 and June 2013, a total of 36 patients received autologous fat grafting in scar areas. Patients who Douleur Neuropathique 4 Questions (scores >4/10) were enrolled this study. The Visual Analogue Scale (VAS), and Neuropathic Pain Symptom Inventory (NPSI) were used to evaluate pain preoperatively and postoperatively after 1 week, 4 weeks, and 24 weeks. The mechanism of trauma, duration of allodynia, fat graft volume, and total follow-up time were recorded.

ELIGIBILITY:
Inclusion Criteria:

* February 2008 and June 2013, patients received autologous fat grafting in scar areas and also had pain over scar area before surgery

Exclusion Criteria:

* patients refused to participate the study

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients received autologous fat grafting in scar areas
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | preoperatively and postoperatively after 1 week, 4 weeks, and 24 weeks.

SECONDARY OUTCOMES:
Neuropathic Pain Symptom Inventory (NPSI) | preoperatively and postoperatively after 1 week, 4 weeks, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: shu-hung huang, MD, Principal Investigator — Division of Plastic Surgery, Department of Surgery, Kaohsiung Medical University Hospital; Chung-Sheng Lai, PhD, Study Chair — Division of Plastic Surgery, Department of Surgery, Kaohsiung Medical University Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan